CLINICAL TRIAL: NCT06402435
Title: A Single-arm, Open, Phase II Clinical Study of SBRT, Chemotherapy, and Ivonescimab Neoadjuvant Therapy for Luminal-type Breast Cancer
Brief Title: SBRT, Chemotherapy, and AK112 Neoadjuvant Therapy for Luminal-type Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Cancer Hospital (Other)
Responsible Party: Principal Investigator, HAN GUANG, professor, Hubei Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBCH-RT-2024-01
Record Dates: First submitted 2024-04-27; First posted 2024-05-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- luminal-type breast cancer patients (Experimental): The study included patients with a histologically confirmed of HR+/HER2-negative (Her2 immunohistochemistry of 0, 1+, or 2+/FISH-) breast cancer who met one of the following criteria: (1) primary tumor mass larger than 2 cm, (2) axillary lymph node metastasis, (3) a willingness to conserve the breasts, but where the ratio of the tumor size to the volume of the breast was large enough to make it difficult to conserve the breasts.
  Interventions: Drug: Lvonescimab (AK112)

INTERVENTIONS:
Drug: Lvonescimab (AK112) — 8Gy×3 SBRT (continuous irradiation) to irradiate the primary lesion (for patients with axillary lymph node metastasis) or 6Gy×3 SBRT (continuous irradiation) to irradiate the primary lesion and axillary lymph node metastasis (for patients without axillary lymph node metastasis) will be administered at first.
  Then the first cycle of chemotherapy + AK112 will be given within 24 hours after the end of SBRT.
  The total eight cycles of preoperative chemotherapy combined with immunotherapy will be administered.
  Surgical resection will be performed within 4-6 weeks after the completion of the eighth cycle.
  The chemotherapy regimen consists of: Four cycles of doxorubicin 50 mg/m² (Q3W) + cyclophosphamide 600 mg/m² (Q3W), followed by Four cycles of albumin-bound paclitaxel 125 mg/m², Day 1 and Day 8 (every 28 days).
  The immunotherapy drug used is Ivonescimab (AK112) (20mg/kg) , administered every 3 weeks concurrently with chemotherapy for 8 cycles.

SUMMARY:
Studies have indicated that the improvement in pathological complete response (pCR) is significantly correlated with luminal breast cancer patients' overall survival (OS). Patients with luminal breast cancer have poor efficacy for neoadjuvant chemotherapy. The combination of neoadjuvant therapy with immunotherapy and chemotherapy has been demonstrated to enhance the pCR rate of luminal-type breast cancer patients, increasing it from 13-15% to approximately 24%. Therefore, how to further improve the pCR rate of luminal-type breast cancer became the main objective of this study. Stereotactic radiotherapy (SBRT) not only kills tumor cells directly, but also kills the distant unirradiated tumor cells by promoting the cross-initiation of tumor-specific CD8+ T cells, a phenomenon known as the abscopal effect. Our research team has recently discovered that the triple therapy model of SBRT + anti-vascular targeting + anti-PD-1 was safe and efficacious in lung cancer patients. Ivonescimab (AK112) is an anti-PD-1/VEGF-A bispecific antibody. In order to improve the pCR, a single-arm, open, phase II clinical study was proposed to explore the safety and efficacy of SBRT+AK112+chemotherapy, a neoadjuvant treatment modality, in the treatment of luminal breast cancer.

ELIGIBILITY:
Inclusion Criteria:

This trial aims to enroll patients who treatment-naïve and voluntarily participate and provide written informed consent; Eligible participants must have histologically confirmed and HR+/HER2-negative breast cancer (HER2 immunohistochemistry 0, 1+, or 2+/FISH-); Patients must meet at least one of the following criteria: (1) tumor size >2 cm, (2) axillary lymph node metastasis, or (3) intent for breast-conserving surgery, but tumor-to-breast volume ratio makes preservation challenging; Additional eligibility requirements include age ≥18 years, an ECOG performance status of 0-1, and baseline laboratory values within acceptable ranges: white blood cell count (WBC) ≥2.0×10⁹/L, absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥100×10⁹/L, hemoglobin (Hb) ≥90 g/L. Liver function parameters must be within ≤1.5×upper limit of normal (ULN) for total bilirubin (TBIL) and ≤3×ULN for alanine aminotransferase (ALT) and aspartate aminotransferase (AST). Renal function must be preserved, with serum creatinine (Cr) ≤1.5× ULN, or if Cr exceeds this limit, the creatinine clearance rate should be ≥50 mL/min (calculated using the Cockcroft-Gault formula). Coagulation parameters should meet the following thresholds: activated partial thromboplastin time (APTT)≤1.5×ULN and prothrombin time (PT) or international normalized ratio (INR) ≤1.5×ULN.

Exclusion Criteria:

Received chemotherapy, targeted therapy, or radiotherapy within 12 months before the first dose of the investigational drug, or have undergone solid organ or hematologic transplantation; A history of myocardial infarction or uncontrolled arrhythmias (QTc ≥470 ms by Fridericia's formula) within 6 months before the first dose; NYHA class III-IV heart failure, left ventricular ejection fraction (LVEF) <50%, or uncontrolled hypertension (systolic BP ≥150 mmHg and/or diastolic BP ≥100 mmHg); Patients with active HIV, tuberculosis, interstitial lung disease, severe pulmonary impairment, or autoimmune diseases requiring systemic immunosuppression will also be excluded; Participants must not have received a live vaccine within 28 days prior to the first dose, though inactivated influenza vaccines are permitted. Patients requiring systemic corticosteroids (>10 mg/day prednisone equivalent) or immunosuppressants within 14 days before the first dose will be excluded, except for short-term or low-dose corticosteroids, localized applications, and adrenal replacement therapy; Patients with active infections requiring systemic therapy within 14 days prior to enrollment, hepatitis B or C with detectable viral DNA/RNA, history of prior treatment with immune checkpoint inhibitors (anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies), participation in another clinical trial within 14 days, major surgery within 4 weeks before the first dose (except for biopsy procedures), severe allergic reactions to monoclonal antibodies or study drug components, pregnancy or lactation, active psychiatric disorders or substance abuse history; Patients who have ceased alcohol consumption may be included. Lastly, investigators may exclude participants based on any other conditions deemed inappropriate for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic remission (pCR) rate | Up to the 30 weeks
  pCR is defined as ypT0/Tis and ypN0

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to the 30 weeks
  Percentage of participants achieving complete response (CR) or partial response (PR), assessed by RECIST v1.1 and iRECIST.
Disease control rate (DCR) | Up to 30 weeks
  Percentage of participants achieving CR, PR, or stable disease (SD), assessed by RECIST v1.1 and iRECIST.
Residual Cancer Burden (RCB) score | At time of surgery
  Quantitative pathological assessment of residual disease in breast and lymph nodes.
Event-free survival (EFS) | Up to 12 months after surgery
  Time from enrollment to disease progression, recurrence, or death.
Safety and tolerability | Through study completion, an average of 1 year after surgery
  Incidence and severity of adverse events graded by CTCAE v5.0.
Quality of life assessment | Pretreatment, Pre-operative, and Up to 12 months after surgery
  Measured using the EORTC QLQ-BR23 and QLQ-C30 questionnaires.

OTHER OUTCOMES:
Minimal residual disease (MRD) dynamics | Up to 12 months after surgery
  MRD assessed at six time points: baseline, after 4 and 8 cycles of neoadjuvant therapy, and at 1, 6, 12 months post-surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei Cancer Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that support the results reported in the publication, including data presented in text, tables, figures, and appendices.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months following publication and ending 3 years after publication.
Access Criteria: 1. With whom will data be shared? Researchers who provide a methodologically sound proposal approved by the study team.
  2. For what types of analyses? For use in individual participant data meta-analyses or other secondary analyses related to breast cancer treatment outcomes.
  3. By what mechanism will data be made available? Upon request via email to the corresponding author, subject to a data use agreement.

REFERENCES:
- [Derived] Zhang C, Bi J, Huang Y, Ke Z, Yuan Z, Ruan H, Pi G, Li Y, Shao J, Han G. Neoadjuvant stereotactic body radiotherapy combined with chemotherapy and Ivonescimab for Chinese luminal-type breast cancer patients: study protocol for a single-arm, open-label, phase II trial. BMJ Open. 2025 Sep 10;15(9):e102952. doi: 10.1136/bmjopen-2025-102952. PMID 40935417